CLINICAL TRIAL: NCT05652751
Title: Effect of Electroacupuncture Combined With NGF on Limb Function in Convalescent Patients With Ischemic Stroke
Brief Title: Effect of EA Combined With NGF on Limb Function in Convalescent Patients With Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Xianming Lin, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Yibinzhao
Record Dates: First submitted 2022-11-30; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke
Keywords: Convalescence; Electroacupuncture; nerve growth factor
MeSH Terms: conditions — Ischemic Stroke; Convalescence; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factor

STUDY DESIGN:
Intervention Model Description: people who are14 days to 6 months after stroke onset
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this trail, it's difficult to blind researchers, because they perform sham EA or EA, and inject NGF or placebo on patients. However, patients, independent outcome assessors and independent statisticians will be blinded to group allocation throughout the entire trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sham EA + placebo group (Placebo Comparator): The sham EA intervention a is that the stimulator is connected to the needle handle on GV20 and GV26 without power for 40 min intervention,once a day for 4 weeks;The patients will receive 1ml volume of physiological saline (PS) injected into the gluteal muscle, once a day for 4 weeks before the sham EA intervention.
  Interventions: Drug: physiological saline; Device: sham EA
- EA + placebo group (Active Comparator): Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle will be inserted in GV20（Baihui) and the stainless needle will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are stimulated by using an acupuncture point nerve stimulator (HANS-200, Nanjing Jinsheng, Ltd., China) with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off), 28 days as a course of treatment, once a day;The patients will receive 1ml volume of physiological saline (PS) injected into the gluteal muscle, once a day for 4 weeks before the EA intervention.
  Interventions: Drug: physiological saline; Device: EA
- sham EA + NGF group (Active Comparator): The sham EA intervention a is that the stimulator is connected to the needle handle on GV20 and GV26 without power for 40 min intervention,once a day for 4 weeks;The 20ug nerve growth factor will be obtained from Hiteck Biopharmaceutical Co., Ltd, Wuhan, China. mNGF will be dissolved in 1 ml sterile water for injection and then injected intramuscularly at gluteal muscle, once a day for 4 weeks before the sham EA intervention. Dose modification is not allowed for mNGF.
  Interventions: Drug: nerve growth factor; Device: sham EA
- EA + NGF group (Active Comparator): Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle will be inserted in GV20（Baihui) and the stainless needle will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness . Then, the needles are stimulated by using an acupuncture point nerve stimulator , 28 days as a course of treatment, once a day;The 20ug nerve growth factor will be dissolved in 1 ml sterile water for injection and then injected intramuscularly at gluteal muscle, once a day for 4 weeks before the EA intervention. Dose modification is not allowed for mNGF.
  Interventions: Drug: nerve growth factor; Device: EA

INTERVENTIONS:
Drug: nerve growth factor — The patient first received an intramuscular injection of NGF or saline into the gluteus maximus.The 20ug nerve growth factor (NO.S20060051, Jinlujie) will be obtained from Hiteck Biopharmaceutical Co., Ltd, Wuhan, China. mNGF will be dissolved in 1 ml sterile water for injection and then injected intramuscularly at gluteal muscle, once a day for 4 weeks. Dose modification is not allowed for mNGF.
  Arms: EA + NGF group; sham EA + NGF group
Drug: physiological saline — Other patients will receive 1ml volume of physiological saline (PS) injected into the gluteal muscle, once a day for 4 weeks.
  Other Names: Sham EA intervention
  Arms: EA + placebo group; sham EA + placebo group
Device: EA — Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle (size 0.25mm×40mm, Hua Tuo brand, Suzhou Medical Supplies Company Ltd in Jiangsu, China) will be inserted in GV20（Baihui) and the stainless needle(size 0.25mm×25mm, described above) will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are stimulated by using an acupuncture point nerve stimulator (HANS-200, Nanjing Jinsheng, Ltd., China) with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off), 28 days as a course of treatment, once a day.
  Arms: EA + NGF group; EA + placebo group
Device: sham EA — The only difference between sham EA intervention and EA intervention is that the stimulator is connected to the needle handle without power for 40 min intervention.
  Arms: sham EA + NGF group; sham EA + placebo group

SUMMARY:
Most ischemic stroke patients are in recovery phase, often accompanied by motor impairment, but they lack effective treatment. The appearance of nerve growth factor (NGF) promotes the development of neuroprotective therapy, but it has little effect on stroke because of the blood-brain barrier (BBB). Electroacupuncture (EA) has been used for stroke, while there is no significant clinical effect for recovery phrase. Consequently, we will conduct a multicentre, randomised, controlled, assessor-blinded clinical trial to assess the effectiveness and safety of EA combined with NGF treatment on ischemic stroke recovery.

ELIGIBILITY:
Inclusion Criteria:

* people with first-ever ischemic stroke confirmed by CT or/and MRI;
* 14 days to 6 months after stroke onset;
* 50 years≤aged≤80 years;
* 3≤modified Rankin Score (mRS)≤4;
* Patients can accept treatment with EA and have good compliance;
* Patients have clear consciousness, pain perception and resolution ability to complete basic communication;
* willing to participate and be randomized to one of the groups.

Exclusion Criteria:

* transient ischemic attack, subarachnoid hemorrhage, cerebral hemorrhage and other cerebrovascular diseases;
* severe heart, liver, kidney dysfunction and severe coagulation dysfunction; cerebral infarction caused by repeated recurrence of stroke, brain surgery or trauma, and brain tumors;
* severe neurological deficits before stroke, such as visual and auditory impairment, aphasia, agnosia, severe hemiplegia, or affected limb function before stroke, such as cerebral palsy, polio, fracture, and mRs≥1;
* diseases with affecting cognitive function such as congenital dementia, or alcohol, drug or substance abuse ;
* lactation, pregnancy or intend to be pregnant within 6 months;
* needlesickness, needle phobia and skin infection at acupuncture site;
* pacemaker, implantable cardioverter defibrillator carriers or conductive metallic foreign bodies in the body;
* allergy to NGF;
* currently enrolled in another clinical trial or participation in other clinical trials within the last 3 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
the modified Rankin Score | the end of treatment (week 4) in all four groups.
  the modified Rankin Score is a common indicator to evaluate motor function in stroke patients.The modified Rankin Score ranges from 0 to 6, and the more severe the neurological deficit, the higher the score.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of motor function score (FMA) | Fugl-Meyer Assessment of motor function score (FMA) is recorded at baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  Fugl-Meyer Assessment of motor function score (FMA) is a common indicator to evaluate motor function.simplified Fugl-Meyer Assessment of motor function score sums up a total score (maximum 100 points ), including an assessment of the upper extremity (maximum 66 points) and lower extremity (maximum 34 points).
Modified Barthel Index (MBI) | Modified Barthel Index (MBI) is recorded at baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  Modified Barthel Index (MBI) is a common indicator to evaluate motor function.The maximum total score of Modified Barthel Index is 100, with a higher score meaning less dependent to help.
timed up and go test (TUGT) | timed up and go test (TUGT) is recorded at baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  timed up and go test (TUGT) is a common indicator to evaluate motor function.In the timed up and go test, each patient is asked to stand up from an armchair at height 45 cm, walk a distance of 3 m, turn, walk back to the chair, and sit back down in chair . With interval of one minute rest, a patient is required to repeat the test three times to take its mean for statistical analysis.
Tinetti Performance Oriented Mobility Assessment (POMA) | Tinetti Performance Oriented Mobility Assessment (POMA) is recorded at baseline (week 0), Mid-term treatment (week 2) and end of treatment (week 4) in all four groups.
  Tinetti Performance Oriented Mobility Assessment (POMA) is a common indicator to evaluate motor function.POMA scale can be used to assess the balance with B-POMA including nine components (sitting balance, arises, attempts to arise, immediate standing balance, standing balance, nudged, eyes closed, turning 360 , and sitting down; maximum 16 points) and to evaluate the gait with G-POMA including seven components (initiation of gait, step length, step symmetry, step continuity, path, trunk, and walking stance; maximum 12 points) . A patient with POMA scored less than 24 points suggets balance dysfunction and scored less than 15 points indicates danger of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No